CLINICAL TRIAL: NCT03992430
Title: A Randomized, Double-Blind, Dose Finding and Comparison Study of the Safety and Efficacy of High Doses of Eteplirsen, Preceded by an Open-label Dose Escalation, in Patients With Duchenne Muscular Dystrophy With Deletion Mutations Amenable to Exon 51 Skipping
Brief Title: A Study to Compare Safety and Efficacy of High Doses of Eteplirsen in Participants With Duchenne Muscular Dystrophy (DMD) (MIS51ON)
Acronym: MIS51ON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4658-402; 2018-001762-42 (EudraCT Number); 2024-511492-15-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne muscular dystrophy; Exon Skipping; Exon 51; North Star Ambulatory Assessment; Ambulatory; DMD; Pediatric; Duchenne; EXONDYS; MIS51ON
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — eteplirsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 is open-label, dose escalation; Part 2 is double-blind, dose finding, and dose comparison
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Eteplirsen (Experimental): Participants will receive eteplirsen 100 mg/kg once weekly for at least 4 weeks, followed by eteplirsen 200 mg/kg once weekly for at least 4 weeks.
  Interventions: Drug: Eteplirsen
- Part 2: Eteplirsen 30 mg/kg (Active Comparator): Randomized participants will receive eteplirsen 30 mg/kg once weekly for up to 144 weeks.
  Interventions: Drug: Eteplirsen
- Part 2: Eteplirsen 100 mg/kg (Experimental): Randomized participants will receive eteplirsen 100 mg/kg once weekly for up to 144 weeks.
  Interventions: Drug: Eteplirsen
- Part 2: Eteplirsen 200 mg/kg (Experimental): Randomized participants will receive eteplirsen 200 mg/kg once weekly for up to 144 weeks.
  Interventions: Drug: Eteplirsen

INTERVENTIONS:
Drug: Eteplirsen — Solution for intravenous (IV) infusion.
  Other Names: AVI-4658; EXONDYS 51; EXONDYS

SUMMARY:
Part 1 (dose escalation) will evaluate the safety and tolerability of 2 doses (100 milligrams/kilogram [mg/kg] and 200 mg/kg) of eteplirsen in approximately 10 participants with DMD; Part 2 (dose finding and dose comparison) will evaluate the efficacy and safety of the high doses (100 mg/kg and 200 mg/kg) of eteplirsen compared with that of the 30 mg/kg dose of eteplirsen, in approximately 144 participants with genetically confirmed deletion mutations amenable to treatment by skipping exon 51.

ELIGIBILITY:
Inclusion Criteria:

* Be a male with an established clinical diagnosis of DMD and an out-of-frame deletion mutation of the DMD gene amenable to exon 51 skipping.
* Ambulatory participant, able to perform TTRISE in 10 seconds or less at the time of screening visit.
* Able to walk independently without assistive devices.
* Have intact right and left biceps muscles or an alternative upper arm muscle group.
* Have been on a stable dose or dose equivalent of oral corticosteroids for at least 12 weeks prior to randomization and the dose is expected to remain constant (except for modifications to accommodate changes in weight and stress-related needs as per the recently published guidelines throughout the study.
* For ages 7 years and older, has stable pulmonary function (forced vital capacity ≥50 percent (%) of predicted and no requirement for nocturnal ventilation). For ages 4 to 6 years, does not require support from ventilator or non-invasive ventilation at time of screening.

Exclusion Criteria:

* Use of any pharmacologic treatment (other than corticosteroids) within 12 weeks prior to randomization.
* Current or previous treatment with any other experimental pharmacologic treatment for DMD or any prior exposure to antisense oligonucleotide, gene therapy or gene editing; except the following: Ezutromid in the last 12 weeks prior to first dose; Drisapersen in the last 36 weeks prior to first dose; Suvodirsen in the last 12 weeks prior to first dose; Vamorolone in the last 12 weeks prior to first dose; Eteplirsen (previous or current use); and Tamoxifen in the last 4 weeks prior to first dose.
* Major surgery within 3 months prior to randomization.
* Presence of any other significant neuromuscular or genetic disease other than DMD.
* Presence of any known impairment of renal function and/or other clinically significant illness.
* Has evidence of cardiomyopathy, as defined by left ventricular ejection fraction less than <50% on the screening echocardiogram or Fridericia's correction formula (QTcF) ≥450 millisecond based on the screening electrocardiograms (ECGs).

Other inclusion/exclusion criteria apply.

Ages: 4 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of Adverse Events (AEs) | Up to Week 148
Part 2: Change From Baseline at Week 144 in the NSAA Total Score (for Final Analysis) | Baseline, Week 144
Part 2: Change from Baseline at Week 72 or Week 96 in NSAA Total Score (for Conditional Efficacy Interim Analysis) | Baseline, Week 72 or Week 96

SECONDARY OUTCOMES:
Part 2: Change From Baseline in Time to Rise From the Floor, Time to Complete 10-Meter Walk/Run, and the Timed Stair Ascend Test | Baseline, Week 144
Part 2: Change From Baseline in the Total Distance Walked During 6-Minute Walk Test (6MWT) | Baseline, Week 144
Part 2: Change from Baseline at Week 144 in Forced Vital Capacity Percent Predicted (FVC%p) | Baseline, Week 144
Part 2: Time to Loss of Ambulation (LOA) | Baseline up to Week 144
Part 2: Change From Baseline in Skeletal Muscle Dystrophin Expression | Baseline, Postdose (at Week 24, Week 48, or Week 144)
Part 2: Incidence of Adverse Events (AEs) | Baseline up to Week 148
Part 2: Pharmacokinetic (PK) Plasma Concentration of Eteplirsen | 0 (predose) to 2 hours postdose up to Week 144

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (59):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida, Gainesville, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá
  - Instituto Neurologico de Colombia (INDEC), Medellín
  - Hospital Pablo Tobón Uribe, Medellín
- Czechia (2):
  - Brno Klinika detske neurologie, Brno
  - Fakultni nemocnice v Motole, Prague
- Rigshospitalet Copenhagen University Hospital, Copenhagen, Denmark
- France (3):
  - Hopital Femme Mere Enfant, Bron
  - Hopital Armand Trousseau, Paris
  - CHRU de Strasbourg, Strasbourg
- Germany (3):
  - Charité Universitätsmedizin Berlin CVK, Berlin
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
- IASO Children's Hospital, Marousi, Attica, Greece
- Semmelweis Egyetem Genomikai Medicina és Ritka Betegsegek Intezete, Budapest, Hungary
- India (8):
  - Royal Institute of Child Neurosciences, Ahmedabad
  - Aster RV Hospital, Bengaluru
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Jaicare Hospital (A Unit of Sarvee Integra Pvt Ltd.), Madurai
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Deenanath Mangeshkar Hospital & Research Centre, Pune
  - Christian Medical College, Vellore
- Children's Health Ireland (CHI) at Temple Street, Dublin, Ireland
- Italy (2):
  - IRCCS Instituto Gianna Gaslini, Genova
  - Fondazione Policlinico Universitario A. Gemelli- IRCCS, Rome
- Jordan (4):
  - The Specialty Hospital (TSH)/Advanced Clinical Center, Amman
  - Istiklal Hosptial (IST), Amman
  - Irbid Specialty Hospital, Irbid
  - Pharmaceutical Research Center/Jordan University of Science and Technology, Irbid
- Mexico (2):
  - Neurociencias Estudios Clínicos S.C., Culiacán, Sinaloa
  - Instituto de Investigaciones Clinicas para la Salud A.C, Durango
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Radboud University Nijmegen Medical Centre, Nijmegen
- New Zealand Clinical Research - Auckland, Auckland, New Zealand
- Norway (2):
  - Oslo Universitetssykehus HF Rikshospitalet, Oslo
  - Children's Department and Department for Children's Habilitation at Stavanger University Hospital, Stavanger
- Klinika Neurologii Rozwojowej, Gdansk, Pomeranian Voivodeship, Poland
- National Clinical Hospital for Children Neurorehabilitation "Dr. Nicolae Robănescu", Bucharest, Romania
- Serbia (3):
  - Clinic for Neurology and Psychiatry for Children and Youth, Belgrade
  - University Children's Hospital, Belgrade
  - Mother and Child Health Care Institute of Serbia "Dr Vukan Cupic", Belgrade
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- South Korea (4):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan
- Spain (2):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Universitätsspital Basel, Basel, Switzerland
- Taiwan (2):
  - Kaohsiung Medical University, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (2):
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Mersin University Medical Faculty, Mersin
- United Kingdom (3):
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire
  - Birmingham Heartlands Hospital, Birmingham
  - UCL Institute of Child Health Great Ormond Street, London